CLINICAL TRIAL: NCT01970137
Title: A 24-week Open-label Study of KPS-0373 in Patients With Spinocerebellar Degeneration (SCD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KPS1304
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Spinocerebellar Degeneration
Keywords: Spinocerebellar degeneration (SCD); Thyrotropin-Releasing Hormone (TRH); Spinocerebellar Ataxia (SCA)
MeSH Terms: conditions — Spinocerebellar Degenerations; Spinocerebellar Ataxias

ARMS (1):
- KPS-0373 (Experimental)
  Interventions: Drug: KPS-0373, High dose; Drug: KPS-0373, Low dose

INTERVENTIONS:
Drug: KPS-0373, High dose
Drug: KPS-0373, Low dose

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and pharmacokinetics of KPS-0373 in SCD patients (Experience of clinical trials of KPS-0373)

ELIGIBILITY:
Inclusion Criteria:

* Japanese SCD patients with ataxia (Experience of clinical trials of KPS-0373)

Exclusion Criteria:

* Patients with secondary ataxia
* Patients with clinically significant hepatic, renal, or cardiovascular dysfunction
* Discontinuations in another clinical trials caused by side effects

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
SARA (Scale for the Assessment and Rating of Ataxia) | 24 weeks

SECONDARY OUTCOMES:
SF-8 (QOL) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo and Other Japanese Cities, Japan